CLINICAL TRIAL: NCT04151628
Title: Prospective, Multicenter, Single-Arm Study of the SWM-1234 in Calcified Coronary Arteries (Disrupt CAD IV Study - Japan)
Brief Title: Disrupt CAD IV With the Shockwave Coronary IVL System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shockwave Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP 62611
Record Dates: First submitted 2019-11-01; First posted 2019-11-05 (Actual); Results first posted 2021-06-25 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2022-04

CONDITIONS: Coronary Artery Disease; Myocardial Infarction
Keywords: Intravascular Lithotripsy; Percutaneous Coronary Intervention
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Infarction | interventions — Lithotripsy

STUDY DESIGN:
Intervention Model Description: The Coronary IVL System is a proprietary balloon catheter system designed to enhance stent outcomes by enabling delivering of the calcium disrupting capability of lithotripsy prior to balloon dilatation at low pressures. The Coronary IVL System consists of an IVL Balloon Catheter with 2 integrated emitters, a Lithotripsy Generator, and a Connector Cable.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Coronary Lithotripsy System (Experimental): All subjects will receive lithotripsy treatment from the Shockwave Medical Coronary IVL System
  Interventions: Device: Lithotripsy

INTERVENTIONS:
Device: Lithotripsy — Deliver Lithotripsy to the target vessel prior to placing a coronary stent

SUMMARY:
The study design is a prospective, multicenter, single-arm study to evaluate the safety and effectiveness of the Shockwave Medical Coronary Intravascular Lithotripsy (IVL) System in de novo, calcified, stenotic coronary arteries prior to stenting.

DETAILED DESCRIPTION:
Subject Population: Subjects ≥ 18 years of age with de novo, calcified coronary artery lesions presenting with stable, unstable or silent ischemia that are suitable for percutaneous coronary intervention. Approximately 72 subjects at 8 sites in Japan will be enrolled. Subjects will be followed through discharge, 30 days, 6, 12 and 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥18 years of age
2. Subjects with native coronary artery disease (including stable or unstable angina and silent ischemia) suitable for PCI
3. For patients with unstable ischemic heart disease, biomarkers (troponin or CK-MB) must be less than or equal to the upper limit of lab normal within 12 hours prior to the procedure (note: if both labs are drawn both must be normal)
4. For patients with stable ischemic heart disease, biomarkers may be drawn prior to the procedure or at the time of the procedure from the side port of the sheath.

   1. If drawn prior to the procedure, biomarkers (troponin or CK- MB) must be less than or equal to the upper limit of lab normal within 12 hours prior to the index procedure (note: if both labs are drawn, both must be normal)
   2. If biomarkers are drawn at the time of the procedure from the side port of the sheath prior to any intervention, biomarker results do not need to be analyzed prior to enrollment.
5. Left ventricular ejection fraction > 25% within 6 months (note: in the case of multiple assessments of LVEF, the measurement closest to enrollment will be used for this criteria; may be assessed at time of index procedure)
6. Subject or legally authorized representative, signs a written Informed Consent form to participate in the study, prior to any study-mandated procedures
7. Lesions in non-target vessels requiring PCI may be treated either:

   1. >30 days prior to the study procedure if the procedure was unsuccessful or complicated; or
   2. >24 hours prior to the study procedure if the procedure was successful and uncomplicated (defined as a final lesion angiographic diameter stenosis <30% and TIMI 3 flow (visually assessed) for all non-target lesions and vessels without perforation, cardiac arrest or need for defibrillation or cardioversion or hypotension/heart failure requiring mechanical or intravenous hemodynamic support or intubation, and with no post-procedure biomarker elevation

      >normal; or
   3. >30 days after the study procedure

   Angiographic Inclusion Criteria
8. The target lesion must be a de novo coronary lesion that has not been previously treated with any interventional procedure
9. Single de novo target lesion stenosis of protected LMCA, or LAD, RCA or LCX (or of their branches) with:

   1. Stenosis of ≥70% and <100% or
   2. Stenosis ≥50% and <70% (visually assessed) with evidence of ischemia via positive stress test, or fractional flow reserve value ≤0.80, or iFR <0.90 or IVUS or OCT minimum lumen area ≤4.0 mm²
10. The target vessel reference diameter must be ≥2.5 mm and ≤4.0 mm
11. The lesion length must not exceed 40 mm
12. The target vessel must have TIMI flow 3 at baseline (visually assessed, may be assessed after pre-dilatation)
13. Evidence of calcification at the lesion site by, a) angiography, with fluoroscopic radio-opacities noted without cardiac motion prior to contrast injection involving both sides of the arterial wall in at least one location and total length of calcium of at least 15 mm and extending partially into the target lesion, OR by b) IVUS or OCT, with presence of ≥270 degrees of calcium on at least 1 cross section
14. Ability to pass a 0.014" guide wire across the lesion

Exclusion Criteria:

1. Any comorbidity or condition which may reduce compliance with this protocol, including follow-up visits
2. Subject is a member of a vulnerable population including individuals with mental disability, persons in nursing homes, children, impoverished persons, persons in emergency situations, homeless persons, nomads, refugees, and those incapable of giving informed consent.
3. Subject is participating in another research study involving an investigational agent (pharmaceutical, biologic, or medical device) that has not reached the primary endpoint
4. Subject is pregnant or nursing (a negative pregnancy test is required for women of child-bearing potential within 7 days prior to enrollment)
5. Unable to tolerate dual antiplatelet therapy (i.e., aspirin, and either clopidogrel, prasugrel, or ticagrelor) for at least 6 months
6. Subject has an allergy to imaging contrast media which cannot be adequately pre-medicated
7. Subject experienced an acute MI (STEMI or non-STEMI) within 30 days prior to index procedure, defined as a clinical syndrome consistent with an acute coronary syndrome with troponin or CK- MB greater than 1 times the local laboratory's upper limit of normal
8. New York Heart Association (NYHA) class III or IV heart failure
9. Renal failure with serum creatinine >2.5 mg/dL, or chronic dialysis
10. History of a stroke or transient ischemic attack (TIA) within 6 months, or any prior intracranial hemorrhage or permanent neurologic deficit
11. Active peptic ulcer or upper gastrointestinal (GI) b≥leeding within 6 months
12. Untreated pre-procedural hemoglobin <10 g/dL or intention to refuse blood transfusions if one should become necessary
13. Coagulopathy, including but not limited to platelet count <100,000 or International Normalized ratio (INR) >1.7 (INR is only required in subjects who have taken warfarin within 2 weeks of enrollment)
14. Subject has a hypercoagulable disorder such as polycythemia vera, platelet count >750,000 or other disorders
15. Uncontrolled diabetes defined as a HbA1c ≥10%
16. Subject has an active systemic infection on the day of the index procedure with either fever, leukocytosis or requiring intravenous antibiotics
17. Subjects in cardiogenic shock or with clinical evidence of left-sided heart failure (S3 gallop, pulmonary rales, oliguria, or hypoxemia)
18. Uncontrolled severe hypertension (systolic BP >180 mm Hg or diastolic BP >110 mm Hg)
19. Subjects with a life expectancy of less than 1 year
20. Non-coronary interventional (e.g., TAVR, MitraClip, or PFO occlusion, etc.) or surgical structural heart procedures within 30 days prior to the index procedure
21. Planned non-coronary interventional (e.g., TAVR, MitraClip, or PFO occlusion, etc.) or surgical structural heart procedures within 30 days after the index procedure
22. Subject refusing or not a candidate for emergency coronary artery bypass grafting (CABG) surgery
23. Planned use of atherectomy, scoring or cutting balloon, or any investigational device other than lithotripsy
24. Unprotected left main diameter stenosis >30%
25. Target vessel is excessively tortuous defined as the presence of two or more bends >90º or three or more bends >75º
26. Definite or possible thrombus (by angiography or intravascular imaging) in the target vessel
27. Evidence of aneurysm in target vessel within 10 mm of the target lesion
28. Target lesion is an ostial location (LAD, LCX, or RCA, within 5 mm of ostium) or an unprotected left main lesion
29. Target lesion is a bifurcation with ostial diameter stenosis ≥30%
30. Second lesion with >50% stenosis in the same target vessel as the target lesion including its side branches
31. Target lesion is located in a native vessel that can only be reached by going through a saphenous vein or arterial bypass graft
32. Previous stent within the target vessel implanted within the last year
33. Previous stent within 10 mm of the target lesion regardless of the timing of its implantation
34. Angiographic evidence of a dissection in the target vessel at baseline or after guidewire passage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2019-11-06 (Actual); Primary Completion 2020-05-08 (Actual); Study Completion 2022-03-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregg W Stone, MD, Study Chair — Columbia University; Shigeru Saito, MD, Principal Investigator — Shonan Kamakura General Hospital
Locations (8):
- Japan (8):
  - Tenjinkai Shin-Koga Hospital, Kurume, Fukuoka
  - Sapporo Higashi Tokushukai Hospital, Sapporo, Hokkaido
  - Sakurakai Takahashi Hospital, Kobe, Hyōgo
  - Higashi-Takarazuka Satoh Hospital, Takarazuka, Hyōgo
  - Shonan-Kamakura General Hospital, Kamakura, Kanagawa
  - Johas Kanto Rosai Hospital, Kawasaki, Kanagawa
  - Kyoto-Katsura Hospital, Kyoto, Kyoto
  - Miyazaki Medical Association Hospital, Miyazaki, Miyazaki

REFERENCES:
- [Result] Saito S, Yamazaki S, Takahashi A, Namiki A, Kawasaki T, Otsuji S, Nakamura S, Shibata Y; Disrupt CAD IV Investigators. Intravascular Lithotripsy for Vessel Preparation in Severely Calcified Coronary Arteries Prior to Stent Placement - Primary Outcomes From the Japanese Disrupt CAD IV Study. Circ J. 2021 May 25;85(6):826-833. doi: 10.1253/circj.CJ-20-1174. Epub 2021 Feb 5. PMID 33551398
- [Derived] Kereiakes DJ, Di Mario C, Riley RF, Fajadet J, Shlofmitz RA, Saito S, Ali ZA, Klein AJ, Price MJ, Hill JM, Stone GW. Intravascular Lithotripsy for Treatment of Calcified Coronary Lesions: Patient-Level Pooled Analysis of the Disrupt CAD Studies. JACC Cardiovasc Interv. 2021 Jun 28;14(12):1337-1348. doi: 10.1016/j.jcin.2021.04.015. Epub 2021 May 3. PMID 33939604

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study enrollment took place at 8 study centers in Japan between November 6, 2019 and April 6, 2020. A total of 72 subjects with de novo, calcified, stenotic coronary arteries were enrolled and treated with the Coronary Intravascular Lithotripsy (IVL) System
Pre-assignment Details: 72 subjects were consented and enrolled into the study
Groups:
- Roll-in: The first subject enrolled at each site is considered a roll-in. Data on roll-in subjects were collected through 30 days, at which time subject participation was complete.
- Intent to Treat (ITT): The Intent to Treat (ITT) population was the primary analysis cohort used to assess the primary safety and effectiveness endpoints. Data on the ITT population was collected through 30 days for primary endpoints. Long-term follow-up for the ITT population to 24 months is complete.
Period: Overall Study
Arm/Group | Roll-in | Intent to Treat (ITT)
Started | 8 | 64
Completed | 8 | 64
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Roll-in | Intent to Treat (ITT) | Total
Number analyzed (Participants) | 8 | 64 | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.3 (3.5) | 75.0 (8.0) | 74.8 (7.7)
Age, Customized [Median (Inter-Quartile Range); unit: years] | 72.5 [70.5 to 76.5] | 74.5 [68.5 to 81.0] | 73.5 [69.0 to 80.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 16 | 18
  Male | 6 | 48 | 54
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 7 | 64 | 71
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 8 | 63 | 71
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Japan | 8 | 64 | 72

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Experienced Freedom From MACE Within 30 Days Post-procedure
Description: The primary safety endpoint was freedom from major adverse cardiac events (MACE) at 30 days - a composite of cardiac death, myocardial infarction (MI) and target vessel revascularization (TVR). The primary endpoints were analyzed using the Intent To Treat (ITT) population.
Time Frame: Within 30 days of index procedure
Population: ITT population was the primary analysis cohort; data on roll-in subjects was only collected through 30 days. Data collected from the roll-in subjects were not pre-specified to be reported as a Primary or Secondary Outcome Measure; therefore, only the ITT arm is reported. The ITT population includes all subjects enrolled in the pivotal phase of the study. This population does not include roll-in subjects.
Measure: Number; unit: percentage of participants
Groups:
- Intent To Treat: The Intent To Treat (ITT) population was the primary analysis cohort used to assess the primary safety and effectiveness endpoints. Data on the ITT population was collected through 30 days for primary endpoints. Long-term follow-up for the ITT population to 24 months is complete.
Arm/Group | Intent To Treat
Number analyzed (Participants) | 64
percentage of participants | 93.8

2. Primary Outcome: Percentage of Subjects With Procedural Success
Description: The primary effectiveness endpoint was Procedural Success defined as stent delivery with a residual in-stent stenosis <50% (core laboratory assessed) and without in-hospital MACE
Time Frame: 12-24 hours post procedure or at discharge, whichever is earlier, but at least 6 hours post procedure
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Intent To Treat
Number analyzed (Participants) | 64
percentage of participants | 93.8

3. Secondary Outcome: Number of Participants With Device Crossing Success
Description: A secondary endpoint was Device Crossing Success defined as the ability to deliver the IVL catheter across the target lesion, and delivery of lithotripsy without serious angiographic complications immediately after IVL. The secondary endpoints were analyzed using the Intent To Treat Analysis Set.
Time Frame: At end of procedure, with a mean total procedure time of 62.5 minutes
Population: Data collected from the roll-in subjects were not pre-specified to be reported as a Secondary Outcome Measure; therefore, only the Intent To Treat group is reported.
Measure: Count of Participants; unit: Participants
Arm/Group | Intent to Treat (ITT)
Number analyzed (Participants) | 64
Participants | 63

4. Secondary Outcome: Number of Participants With Angiographic Success (Residual Stenosis <50%)
Description: A secondary endpoint was Angiographic Success defined as stent delivery with <50%residual stenosis and without serious angiographic complications. The secondary endpoints were analyzed using the Intent To Treat Analysis Set.
Time Frame: At end of procedure, with a mean total procedure time of 62.5 minutes
Population: Data collected from the roll-in subjects were not pre-specified to be reported as a Secondary Outcome Measure; therefore, only the Intent To Treat population is reported.
Measure: Count of Participants; unit: Participants
Arm/Group | Intent to Treat (ITT)
Number analyzed (Participants) | 64
Participants | 63

5. Secondary Outcome: Number of Participants With Procedural Success (Residual Stenosis <=30%)
Description: secondary endpoint was Procedural Success defined as stent delivery with aresidual stenosis <=30% (core laboratory assessed) and without in-hospital MACE. The secondary endpoints were analyzed using the Intent To Treat Analysis Set.
Time Frame: 12-24 hours post procedure or at discharge, whichever is earlier, but at least 6 hours post procedure
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Intent to Treat (ITT)
Number analyzed (Participants) | 64
Participants | 60

6. Secondary Outcome: Number of Participants With Angiographic Success (Residual Stenosis <=30%)
Description: A secondary endpoint was Angiographic Success defined as stent delivery with<=30% residual stenosis and without serious angiographic complications. These secondary endpoints were analyzed using the Intent To Treat Analysis Set.
Time Frame: At end of procedure, with a mean total procedure time of 62.5 minutes
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Intent to Treat (ITT)
Number analyzed (Participants) | 64
Participants | 63

7. Secondary Outcome: Number of Participants With Serious Angiographic Complications
Description: A secondary endpoint was Serious Angiographic Complications defined as severedissection (Type D to F), perforation, abrupt closure, and persistent slow flow or persistent no reflow. The secondary endpoints were analyzed using the Intent To Treat Analysis Set.
Time Frame: At end of procedure, with a mean total procedure time of 62.5 minutes
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Intent to Treat (ITT)
Number analyzed (Participants) | 64
Participants | 63

8. Secondary Outcome: MACE Rate at 6 Months
Description: The MACE rate at 6 months - a composite of cardiac death, myocardial infarction (MI) and target vessel revascularization (TVR)- is presented as Kaplan-Meier (K-M) estimated event rate. The secondary endpoints were analyzed using the Intent To Treat Analysis Set.
Time Frame: within 6 months of index procedure
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Intent to Treat (ITT)
Number analyzed (Participants) | 64
percentage of participants | 7.8

9. Secondary Outcome: MACE Rate at 12 Months
Description: The MACE rate at 12 months - a composite of cardiac death, myocardial infarction (MI) and target vessel revascularization (TVR)- is presented as Kaplan-Meier (K-M) estimated event rate. The secondary endpoints were analyzed using the Intent To Treat Analysis Set.
Time Frame: within 12 months of index procedure
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Intent to Treat (ITT)
Number analyzed (Participants) | 64
percentage of participants | 9.4

10. Secondary Outcome: MACE Rate at 24 Months
Description: The MACE rate at 24 months - a composite of cardiac death, myocardial infarction (MI) and target vessel revascularization (TVR)- is presented as Kaplan-Meier (K-M) estimated event rate. The secondary endpoints were analyzed using the Intent To Treat Analysis Set.
Time Frame: within 24 months of index procedure
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Intent to Treat (ITT)
Number analyzed (Participants) | 64
percentage of participants | 12.6

11. Secondary Outcome: Target Lesion Failure (TLF) at 30 Days
Description: Target Lesion Failure (TLF) is defined as cardiac death, target vessel MI (TV-MI) or ischemia-driven target lesion revascularization (ID-TLR), and is presented as proportions at 30 days. The secondary endpoints were analyzed using the Intent To Treat Analysis Set.
Time Frame: Within 30 days of index procedure
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Intent to Treat (ITT)
Number analyzed (Participants) | 64
percentage of participants | 6.3

12. Secondary Outcome: Target Lesion Failure (TLF) at 6 Months
Description: Target Lesion Failure (TLF) is defined as cardiac death, target vessel MI (TV-MI) or ischemia-driven target lesion revascularization (ID-TLR). TLF is presented as Kaplan-Meier estimated event rate at 6 months. The secondary endpoints were analyzed using the Intent To Treat Analysis Set.
Time Frame: Within 6 months of index procedure
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Intent to Treat (ITT)
Number analyzed (Participants) | 64
percentage of participants | 6.3

13. Secondary Outcome: Target Lesion Failure (TLF) at 12 Months
Description: Target Lesion Failure (TLF) is defined as cardiac death, target vessel MI (TV-MI) or ischemia-driven target lesion revascularization (ID-TLR). TLF is presented as Kaplan-Meier estimated event rate at 12 months. The secondary endpoints were analyzed using the Intent To Treat Analysis Set.
Time Frame: Within 12 months of index procedure
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Intent to Treat (ITT)
Number analyzed (Participants) | 64
percentage of participants | 6.3

14. Secondary Outcome: Target Lesion Failure (TLF) at 24 Months
Description: Target Lesion Failure (TLF) is defined as cardiac death, target vessel MI (TV-MI) or ischemia-driven target lesion revascularization (ID-TLR). TLF is presented as Kaplan-Meier estimated event rate at 24 months. The secondary endpoints were analyzed using the Intent To Treat Analysis Set.
Time Frame: Within 24 months of index procedure
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Intent to Treat (ITT)
Number analyzed (Participants) | 64
percentage of participants | 7.8

15. Secondary Outcome: All-Cause Death at 30 Days
Description: The 30-day rates of all-cause death are presented as proportions. The secondary endpoints were analyzed using the Intent To Treat Analysis Set.
Time Frame: Within 30 days from index procedure
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Intent to Treat (ITT)
Number analyzed (Participants) | 64
percentage of participants | 0

16. Secondary Outcome: All-Cause Death at 6 Months
Description: All-cause death at 6 months is presented as Kaplan-Meier estimated event rate. The secondary endpoints were analyzed using the Intent To Treat Analysis Set.
Time Frame: within 6 months of index procedure
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Intent to Treat (ITT)
Number analyzed (Participants) | 64
percentage of participants | 0

17. Secondary Outcome: All-Cause Death at 12 Months
Description: All-cause death at 12 month is presented as Kaplan-Meier estimated event rate. The secondary endpoints were analyzed using the Intent To Treat Analysis Set.
Time Frame: within 12 months of procedure
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Intent to Treat (ITT)
Number analyzed (Participants) | 64
percentage of participants | 0

18. Secondary Outcome: All-Cause Death at 24 Months
Description: All-cause death at 24 month is presented as Kaplan-Meier estimated event rate. The secondary endpoints were analyzed using the Intent To Treat Analysis Set.
Time Frame: within 24 months of procedure
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Intent to Treat (ITT)
Number analyzed (Participants) | 64
percentage of participants | 3.1

19. Secondary Outcome: Myocardial Infarction (MI) at 30 Days
Description: The 30-day MI rates are presented as proportions. The secondary endpoints were analyzed using the Intent To Treat Analysis Set.
Time Frame: within 30 days of index procedure
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Intent to Treat (ITT)
Number analyzed (Participants) | 64
percentage of participants | 6.3

20. Secondary Outcome: Myocardial Infarction (MI) at 6 Months
Description: MI is presented as Kaplan-Meier estimated event rate at 6 months. The secondary endpoints were analyzed using the Intent To Treat Analysis Set.
Time Frame: Within 6 months of index procedure
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Intent to Treat (ITT)
Number analyzed (Participants) | 64
percentage of participants | 6.3

21. Secondary Outcome: Myocardial Infarction (MI) at 12 Months
Description: MI is presented as Kaplan-Meier estimated event rate at 12 months. The secondary endpoints were analyzed using the Intent To Treat Analysis Set.
Time Frame: Within 12 months of index procedure
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Intent to Treat (ITT)
Number analyzed (Participants) | 64
percentage of participants | 6.3

22. Secondary Outcome: Myocardial Infarction (MI) at 24 Months
Description: MI is presented as Kaplan-Meier estimated event rate at 24 months. The secondary endpoints were analyzed using the Intent To Treat Analysis Set.
Time Frame: Within 24 months of index procedure
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Intent to Treat (ITT)
Number analyzed (Participants) | 64
percentage of participants | 6.3

23. Secondary Outcome: Myocardial Infarction Attributable to Target Vessel (TV-MI) at 30 Days
Description: The Myocardial Infarction attributable to the target vessel (TV-MI) rates at 30 days are presented as proportions. The secondary endpoints were analyzed using the Intent To Treat Analysis Set.
Time Frame: within 30 days of index procedure
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Intent to Treat (ITT)
Number analyzed (Participants) | 64
percentage of participants | 6.3

24. Secondary Outcome: Myocardial Infarction Attributable to Target Vessel (TV-MI) at 6 Months
Description: The Myocardial Infarction attributable to the target vessel (TV-MI) is presented as Kaplan-Meier estimated event rate at 6 months. The secondary endpoints were analyzed using the Intent To Treat Analysis Set.
Time Frame: Within 6 month of index procedure
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Intent to Treat (ITT)
Number analyzed (Participants) | 64
percentage of participants | 6.3

25. Secondary Outcome: Myocardial Infarction Attributable to Target Vessel (TV-MI) at 12 Months
Description: The Myocardial Infarction attributable to the target vessel (TV-MI) is presented as Kaplan-Meier estimated event rate at 12 months. The secondary endpoints were analyzed using the Intent To Treat Analysis Set.
Time Frame: Within 12 months of index procedure
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Intent to Treat (ITT)
Number analyzed (Participants) | 64
percentage of participants | 6.3

26. Secondary Outcome: Myocardial Infarction Attributable to Target Vessel (TV-MI) at 24 Months
Description: The Myocardial Infarction attributable to the target vessel (TV-MI) is presented as Kaplan-Meier estimated event rate at 24 months. The secondary endpoints were analyzed using the Intent To Treat Analysis Set.
Time Frame: Within 24 months of index procedure
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Intent to Treat (ITT)
Number analyzed (Participants) | 64
percentage of participants | 6.3

27. Secondary Outcome: Stent Thrombosis at 30 Days
Description: The Stent Thrombosis rate at 30 days is presented as a proportion. The secondary endpoints were analyzed using the Intent To Treat Analysis Set.
Time Frame: Within 30 days of index procedure
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Intent to Treat (ITT)
Number analyzed (Participants) | 64
percentage of participants | 0

28. Secondary Outcome: Stent Thrombosis at 6 Months
Description: Stent thrombosis is presented as Kaplan-Meier estimated event rate at 6 months. The secondary endpoints were analyzed using the Intent To Treat Analysis Set.
Time Frame: within 6 months of index procedure
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Intent to Treat (ITT)
Number analyzed (Participants) | 64
percentage of participants | 0

29. Secondary Outcome: Stent Thrombosis at 12 Months
Description: Stent thrombosis is presented as Kaplan-Meier estimated event rate at 12 months. The secondary endpoints were analyzed using the Intent To Treat Analysis Set.
Time Frame: within 12 months of index procedure
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Intent to Treat (ITT)
Number analyzed (Participants) | 64
percentage of participants | 0

30. Secondary Outcome: Stent Thrombosis at 24 Months
Description: Stent thrombosis is presented as Kaplan-Meier estimated event rate at 24 months. The secondary endpoints were analyzed using the Intent To Treat Analysis Set.
Time Frame: within 24 months of index procedure
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Intent to Treat (ITT)
Number analyzed (Participants) | 64
percentage of participants | 0

31. Secondary Outcome: All Revascularizations at 30 Days
Description: The 30-day revascularization rate is presented as a proportion. The secondary endpoints were analyzed using the Intent To Treat Analysis Set.
Time Frame: within 30 days of index procedure
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Intent To Treat
Number analyzed (Participants) | 64
percentage of participants | 0

32. Secondary Outcome: All Revascularizations at 6 Months
Description: All revascularizations are presented as Kaplan-Meier estimated event rates at 6 months. The secondary endpoints were analyzed using the Intent To Treat Analysis Set.
Time Frame: within 6 months of index procedure
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Intent To Treat
Number analyzed (Participants) | 64
percentage of participants | 12.5

33. Secondary Outcome: All Revascularizations at 12 Months
Description: All revascularizations are presented as Kaplan-Meier estimated event rates at 12 months. The secondary endpoints were analyzed using the Intent To Treat Analysis Set.
Time Frame: within 12 months of index procedure
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Intent To Treat
Number analyzed (Participants) | 64
percentage of participants | 15.6

34. Secondary Outcome: All Revascularizations at 24 Months
Description: All revascularizations are presented as Kaplan-Meier estimated event rates at 24 months. The secondary endpoints were analyzed using the Intent To Treat Analysis Set.
Time Frame: within 24 months of index procedure
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Intent to Treat (ITT)
Number analyzed (Participants) | 64
percentage of participants | 20.4

35. Secondary Outcome: Ischemia-Driven Target Vessel Revascularization (ID-TVR) at 30 Days
Description: The ischemia-driven Target Vessel Revascularization at 30 days is presented as a proportion. The secondary endpoints were analyzed using the Intent To Treat Analysis Set.
Time Frame: within 30 days of index procedure
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Intent To Treat
Number analyzed (Participants) | 64
percentage of participants | 0

36. Secondary Outcome: Ischemia-Driven Target Vessel Revascularization (ID-TVR) at 6 Months
Description: The ischemia-driven Target Vessel Revascularization (ID-TVR) is presented as Kaplan-Meier estimated event rate at 6 months. The secondary endpoints were analyzed using the Intent To Treat Analysis Set.
Time Frame: within 6 months of index procedure
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Intent To Treat
Number analyzed (Participants) | 64
percentage of participants | 3.1

37. Secondary Outcome: Ischemia-driven Target Vessel Revascularization (ID-TVR) at 12 Months
Description: The ischemia-driven Target Vessel Revascularization (ID-TVR) is presented as Kaplan-Meier estimated event rate at 12 months. The secondary endpoints were analyzed using the Intent To Treat Analysis Set.
Time Frame: within 12 months of index procedure
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Intent To Treat
Number analyzed (Participants) | 64
percentage of participants | 4.7

38. Secondary Outcome: Ischemia-driven Target Vessel Revascularization (ID-TVR) at 24 Months
Description: The ischemia-driven Target Vessel Revascularization (ID-TVR) is presented as Kaplan-Meier estimated event rate at 24 months. The secondary endpoints were analyzed using the Intent To Treat Analysis Set.
Time Frame: within 24 months of index procedure
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Intent to Treat (ITT)
Number analyzed (Participants) | 64
percentage of participants | 7.9

39. Secondary Outcome: Ischemia-Driven Target Lesion Revascularization (ID-TLR) at 30 Days
Description: The ischemia-driven Target Lesion Revascularization (ID-TLR) 30-day rate is presented as a proportion. The secondary endpoints were analyzed using the Intent To Treat Analysis Set.
Time Frame: within 30 days of index procedure
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Intent To Treat
Number analyzed (Participants) | 64
percentage of participants | 0

40. Secondary Outcome: Ischemia-Driven Target Lesion Revascularization (ID-TLR) at 6 Months
Description: The ischemia-driven Target Lesion Revascularization (ID-TLR) is presented as Kaplan-Meier estimated event rate at 6 months. The secondary endpoints were analyzed using the Intent To Treat Analysis Set.
Time Frame: within 6 months of index procedure
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Intent To Treat
Number analyzed (Participants) | 64
percentage of participants | 1.6

41. Secondary Outcome: Ischemia-Driven Target Lesion Revascularization (ID-TLR) at 12 Months
Description: The ischemia-driven Target Lesion Revascularization (ID-TLR) is presented as Kaplan-Meier estimated event rate at 12 months. The secondary endpoints were analyzed using the Intent To Treat Analysis Set.
Time Frame: within 12 months of index procedure
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Intent To Treat
Number analyzed (Participants) | 64
percentage of participants | 1.6

42. Secondary Outcome: Ischemia-Driven Target Lesion Revascularization (ID-TLR) at 24 Months
Description: The ischemia-driven Target Lesion Revascularization (ID-TLR) is presented as Kaplan-Meier estimated event rate at 24 months. The secondary endpoints were analyzed using the Intent To Treat Analysis Set.
Time Frame: within 24 months of index procedure
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Intent to Treat (ITT)
Number analyzed (Participants) | 64
percentage of participants | 3.2

43. Secondary Outcome: Non-Ischemia-Driven Target Vessel Revascularization (Non-ID-TVR) at 30 Days
Description: The non-ischemia-driven Target Vessel Revascularization (Non-ID-TVR) 30-day rate is presented as a proportion. The secondary endpoints were analyzed using the Intent To Treat Analysis Set.
Time Frame: within 30 days of index procedure
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Intent To Treat
Number analyzed (Participants) | 64
percentage of participants | 0

44. Secondary Outcome: Non-Ischemia-Driven Target Vessel Revascularization (Non-ID-TVR) at 6 Months
Description: The non-ischemia-driven Target Vessel Revascularization (Non-ID-TVR) is presented as Kaplan-Meier estimated event rate at 6 months. The secondary endpoints were analyzed using the Intent To Treat Analysis Set.
Time Frame: within 6 months of index procedure
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Intent To Treat
Number analyzed (Participants) | 64
percentage of participants | 0

45. Secondary Outcome: Non-Ischemia-Driven Target Vessel Revascularization (Non-ID-TVR) at 12 Months
Description: The non-ischemia-driven Target Vessel Revascularization (Non-ID-TVR) is presented as Kaplan-Meier estimated event rate at 12 months. The secondary endpoints were analyzed using the Intent To Treat Analysis Set.
Time Frame: within 12 months of index procedure
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Intent To Treat
Number analyzed (Participants) | 64
percentage of participants | 0

46. Secondary Outcome: Non-Ischemia-Driven Target Vessel Revascularization (Non-ID-TVR) at 24 Months
Description: The non-ischemia-driven Target Vessel Revascularization (Non-ID-TVR) is presented as Kaplan-Meier estimated event rate at 24 months. The secondary endpoints were analyzed using the Intent To Treat Analysis Set.
Time Frame: within 24 months of index procedure
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Intent to Treat (ITT)
Number analyzed (Participants) | 64
percentage of participants | 0

47. Secondary Outcome: Non-Ischemia-Driven Target Lesion Revascularization (Non-ID-TLR) at 30 Days
Description: The non-ischemia-driven Target Lesion Revascularization (Non-ID-TLR) 30-day rate is presented as a proportion. The secondary endpoints were analyzed using the Intent To Treat Analysis Set.
Time Frame: within 30 days of index procedure
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Intent To Treat
Number analyzed (Participants) | 64
percentage of participants | 0

48. Secondary Outcome: Non-Ischemia-Driven Target Lesion Revascularization (Non-ID-TLR) at 6 Months
Description: The non-ischemia-driven Target Lesion Revascularization (Non-ID-TLR) is presented as Kaplan-Meier estimated event rate at 6 months. The secondary endpoints were analyzed using the Intent To Treat Analysis Set.
Time Frame: within 6 months of index procedure
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Intent To Treat
Number analyzed (Participants) | 64
percentage of participants | 0

49. Secondary Outcome: Non-Ischemia-Driven Target Lesion Revascularization (Non-ID-TLR) at 12 Months
Description: The non-ischemia-driven Target Lesion Revascularization (Non-ID-TLR) is presented as Kaplan-Meier estimated event rate at 12 months. The secondary endpoints were analyzed using the Intent To Treat Analysis Set.
Time Frame: within 12 months of index procedure
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Intent To Treat
Number analyzed (Participants) | 64
percentage of participants | 0

50. Secondary Outcome: Non-Ischemia-Driven Target Lesion Revascularization (Non-ID-TLR) at 24 Months
Description: The non-ischemia-driven Target Lesion Revascularization (Non-ID-TLR) is presented as Kaplan-Meier estimated event rate at 24 months. The secondary endpoints were analyzed using the Intent To Treat Analysis Set.
Time Frame: within 24 months of index procedure
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Intent to Treat (ITT)
Number analyzed (Participants) | 64
percentage of participants | 0

51. Secondary Outcome: Procedural MI at 30 Days
Description: The procedural MI 30-day rate is presented as a proportion. The secondary endpoints were analyzed using the Intent To Treat Analysis Set.
Time Frame: within 30 days of index procedure
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Intent To Treat
Number analyzed (Participants) | 64
percentage of participants | 6.3

52. Secondary Outcome: Procedural MI at 6 Months
Description: The procedural MI is presented as Kaplan-Meier estimated event rate at 6 months. The secondary endpoints were analyzed using the Intent To Treat Analysis Set.
Time Frame: within 6 months of index procedure
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Intent To Treat
Number analyzed (Participants) | 64
percentage of participants | 6.3

53. Secondary Outcome: Procedural MI at 12 Months
Description: The procedural MI is presented as Kaplan-Meier estimated event rate at 12 months. The secondary endpoints were analyzed using the Intent To Treat Analysis Set.
Time Frame: within 12 months of index procedure
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Intent To Treat
Number analyzed (Participants) | 64
percentage of participants | 6.3

54. Secondary Outcome: Procedural MI at 24 Months
Description: The procedural MI is presented as Kaplan-Meier estimated event rate at 24 months. The secondary endpoints were analyzed using the Intent To Treat Analysis Set.
Time Frame: within 24 months of index procedure
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Intent to Treat (ITT)
Number analyzed (Participants) | 64
percentage of participants | 6.3

55. Secondary Outcome: Non-Procedural MI at 30 Days
Description: The non-procedural MI 30-day rate is presented as a proportion. The secondary endpoints were analyzed using the Intent To Treat Analysis Set.
Time Frame: within 30 days of index procedure
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Intent To Treat
Number analyzed (Participants) | 64
percentage of participants | 0

56. Secondary Outcome: Non-Procedural MI at 6 Months
Description: The non-procedural MI is presented as Kaplan-Meier estimated event rate at 6 months. The secondary endpoints were analyzed using the Intent To Treat Analysis Set.
Time Frame: within 6 months of index procedure
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Intent To Treat
Number analyzed (Participants) | 64
percentage of participants | 0

57. Secondary Outcome: Non-Procedural MI at 12 Months
Description: The non-procedural MI is presented as Kaplan-Meier estimated event rate at 12 months. The secondary endpoints were analyzed using the Intent To Treat Analysis Set.
Time Frame: within 12 months of index procedure
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Intent To Treat
Number analyzed (Participants) | 64
percentage of participants | 0

58. Secondary Outcome: Non-Procedural MI at 24 Months
Description: The non-procedural MI is presented as Kaplan-Meier estimated event rate at 24 months. The secondary endpoints were analyzed using the Intent To Treat Analysis Set.
Time Frame: within 24 months of index procedure
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Intent to Treat (ITT)
Number analyzed (Participants) | 64
percentage of participants | 0

59. Secondary Outcome: Myocardial Infarction (MI) Using the Fourth Universal Definition of MI, at 30 Days
Description: The 30-day rate of MI using the Fourth Universal Definition of MI is presented as a proportion. The secondary endpoints were analyzed using the Intent To Treat Analysis Set.
Time Frame: within 30 days of index procedure
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Intent To Treat
Number analyzed (Participants) | 64
percentage of participants | 7.8

60. Secondary Outcome: Myocardial Infarction (MI) Using the Fourth Universal Definition of MI, at 6 Months
Description: MI using the Fourth Universal Definition of MI is presented as Kaplan-Meier estimated event rate at 6 months. The secondary endpoints were analyzed using the Intent To Treat Analysis Set.
Time Frame: within 6 months of index procedure
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Intent To Treat
Number analyzed (Participants) | 64
percentage of participants | 7.8

61. Secondary Outcome: Myocardial Infarction (MI) Using the Fourth Universal Definition of MI, at 12 Months
Description: MI using the Fourth Universal Definition of MI is presented as Kaplan-Meier estimated event rate at 12 months. The secondary endpoints were analyzed using the Intent To Treat Analysis Set.
Time Frame: within 12 months of index procedure
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Intent To Treat
Number analyzed (Participants) | 64
percentage of participants | 7.8

62. Secondary Outcome: Myocardial Infarction (MI) Using the Fourth Universal Definition of MI, at 24 Months
Description: MI using the Fourth Universal Definition of MI is presented as Kaplan-Meier estimated event rate at 24 months. The secondary endpoints were analyzed using the Intent To Treat Analysis Set.
Time Frame: within 24 months of index procedure
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Intent to Treat (ITT)
Number analyzed (Participants) | 64
percentage of participants | 7.8

63. Secondary Outcome: Myocardial Infarction (MI) Using the Society for Cardiovascular Angiography and Interventions (SCAI) Definition, at 30 Days
Description: The 30-day rate of MI using the SCAI Definition of MI is presented as a proportion. The secondary endpoints were analyzed using the Intent To Treat Analysis Set.
Time Frame: within 30 days of index procedure
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Intent To Treat
Number analyzed (Participants) | 64
percentage of participants | 3.1

64. Secondary Outcome: Myocardial Infarction (MI) Using the Society for Cardiovascular Angiography and Interventions (SCAI) Definition, at 6 Months
Description: MI using the SCAI definition is presented as Kaplan-Meier estimated event rate at 6 months. The secondary endpoints were analyzed using the Intent To Treat Analysis Set.
Time Frame: within 6 months of index procedure
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Intent To Treat
Number analyzed (Participants) | 64
percentage of participants | 3.1

65. Secondary Outcome: Myocardial Infarction (MI) Using the Society for Cardiovascular Angiography and Interventions (SCAI) Definition, at 12 Months
Description: MI using the SCAI definition is presented as Kaplan-Meier estimated event rate at 12 months. The secondary endpoints were analyzed using the Intent To Treat Analysis Set.
Time Frame: within 12 months of index procedure
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Intent To Treat
Number analyzed (Participants) | 64
percentage of participants | 3.1

66. Secondary Outcome: Myocardial Infarction (MI) Using the Society for Cardiovascular Angiography and Interventions (SCAI) Definition, at 24 Months
Description: MI using the SCAI definition is presented as Kaplan-Meier estimated event rate at 24 months. The secondary endpoints were analyzed using the Intent To Treat Analysis Set.
Time Frame: within 24 months of index procedure
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Intent to Treat (ITT)
Number analyzed (Participants) | 64
percentage of participants | 3.1

ADVERSE EVENTS:
Time Frame: within 30 days of index procedure for both Roll-In and Intent To Treat arms, and through 24 months for Intent To Treat arm only
Groups:
- Coronary IVL System(Roll-In) Through 30Days: Adverse events reported through 30 days post-procedure for Roll-In subjects. The first subject enrolled at each site is considered a roll-in. Per protocol, data on roll-in subjects were collected through 30days, at which time subject participation was complete.
- Coronary IVL System(ITT) Through 30Days: Adverse events reported through 30 days post-procedure for ITT subjects. The ITT analysis set was the primary analysis cohort used to assess the primary safety and effectiveness endpoints.
- Coronary IVL System(ITT) Through 12Months: Adverse events reported through 12 months post-procedure for ITT subjects. Adverse event data on ITT subjects was collected through12 months for long-term follow-up. Long-term follow-up for ITT subjects to 24 months is complete.
- Coronary IVL System (ITT) Through 24 Months: Adverse events reported through 24 months post-procedure for ITT subjects. Adverse event data on ITT subjects was collected through 24 months for long-term follow-up. Long-term follow-up for ITT subjects to 24 months is complete.
Arm/Group | Coronary IVL System(Roll-In) Through 30Days | Coronary IVL System(ITT) Through 30Days | Coronary IVL System(ITT) Through 12Months | Coronary IVL System (ITT) Through 24 Months
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/64 | 0/64 | 2/64
Serious Adverse Events (participants affected / at risk) | 0/8 | 5/64 | 23/64 | 30/64
Other Adverse Events (participants affected / at risk) | 1/8 | 11/64 | 14/64 | 14/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Coronary IVL System(Roll-In) Through 30Days (N=8) | Coronary IVL System(ITT) Through 30Days (N=64) | Coronary IVL System(ITT) Through 12Months (N=64) | Coronary IVL System (ITT) Through 24 Months (N=64)
Coronary Artery Occlusion (Cardiac disorders) | 0 | 1 (1) | 1 (1) | 2 (2)
Myocardial Infarction (Cardiac disorders) | 0 | 1 (1) | 1 (1) | 1 (1)
Retroperitoneal Mass (Gastrointestinal disorders) | 0 | 1 (1) | 1 (1) | 1 (1)
Periodontitis (Infections and infestations) | 0 | 1 (1) | 1 (1) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 | 1 (1) | 2 (2) | 3 (3)
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1 (1) | 2 (2) | 2 (2)
Myocardial ischemia (Cardiac disorders) | 0 | 0 | 2 (2) | 2 (2)
Angina Pectoris (Cardiac disorders) | 0 | 0 | 1 (1) | 2 (2)
Angina unstable (Cardiac disorders) | 0 | 0 | 1 (1) | 1 (1)
Arrhythmia (Cardiac disorders) | 0 | 0 | 1 (1) | 2 (2)
Cardiac Failure Congestive (Cardiac disorders) | 0 | 0 | 1 (1) | 2 (2)
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 2 (2) | 2 (2)
Large Intestine Polyp (Gastrointestinal disorders) | 0 | 0 | 1 (1) | 1 (1)
Mechanical ileus (Gastrointestinal disorders) | 0 | 0 | 1 (1) | 1 (2)
Oedema peripheral (General disorders) | 0 | 0 | 1 (1) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 2 (3) | 2 (3)
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 1 (1) | 1 (2)
Jaundice (Hepatobiliary disorders) | 0 | 0 | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 0 | 0 | 1 (1) | 1 (1)
Infected dermal cyst (Infections and infestations) | 0 | 0 | 1 (1) | 1 (1)
Pelvic abscess (Infections and infestations) | 0 | 0 | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 0 | 0 | 1 (1) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 (1) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 (1) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 (1) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 (1) | 1 (1)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 (1) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 (1) | 1 (1)
Pancreatic neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 (1) | 1 (1)
Haemorrhage (Vascular disorders) | 0 | 0 | 2 (2) | 2 (2)
Aortic stenosis (Vascular disorders) | 0 | 0 | 1 (1) | 1 (1)
Peripheral ischemia (Vascular disorders) | 0 | 0 | 1 (1) | 1 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Coronary IVL System(Roll-In) Through 30Days (N=8) | Coronary IVL System(ITT) Through 30Days (N=64) | Coronary IVL System(ITT) Through 12Months (N=64) | Coronary IVL System (ITT) Through 24 Months (N=64)
Coronary artery dissection (Cardiac disorders) | 0 | 11 (11) | 12 (12) | 12 (12) — Roll-In group does not meet 5% frequency threshold for reporting
Vascular Access Site Complication (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 2 (2) | 2 (2) — ITT group does not meet 5% frequency threshold for reporting
Hypotension (Vascular disorders) | 1 (1) | 2 (2) | 2 (2) | 2 (2) — ITT group does not meet 5% frequency threshold for reporting
Constipation (Gastrointestinal disorders) | 0 | 1 (1) | 4 (4) | 4 (4) — Roll-In and ITT groups do not meet the 5% frequency threshold for reporting

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-19): https://cdn.clinicaltrials.gov/large-docs/28/NCT04151628/Prot_SAP_001.pdf